CLINICAL TRIAL: NCT00795301
Title: A Randomized, Phase II Study of Concurrent Radiotherapy and Oxaliplatin, Capecitabine With or Without Cetuximab in Rectal Cancer Tumor Stratified by KRAS Mutation Status.
Brief Title: A Study of Radiotherapy in Rectal Cancer Using Oxaliplatin, Capecitabine With or Without Cetuximab
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Wei Peng Yong, National University Hospital
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CR02/06/07
Record Dates: First submitted 2008-11-20; First posted 2008-11-21 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2014-01

CONDITIONS: Rectal Cancer
Keywords: tumor
MeSH Terms: conditions — Rectal Neoplasms; Neoplasms | interventions — Capecitabine; Cetuximab; Oxaliplatin

INTERVENTIONS:
Drug: Capecitabine, Cetuximab, Oxaliplatin

SUMMARY:
Primary Objectives To estimate the pathological complete response rate following neoadjuvant radiotherapy with concurrent capecitabine and oxaliplatin, with or without cetuximab based on the KRAS mutation status in rectal cancer.

Secondary Objectives

1. To evaluate the incidence of grade 3-4 toxicities with each of the two neoadjuvant regimens and during the 30-day post-operative period.
2. To estimate the clinical tumour response rate and sphincter preservation rate with each of the two neoadjuvant regimens.
3. To correlate EGRF gene amplification with pathological response rate in those treated with cetuximab.
4. To estimate the pattern of failure.
5. To establish an annotated tissue library with samples being obtained prior to therapy and following therapy (at the time of surgery).

DETAILED DESCRIPTION:
Aims: The primary aim of this study is to estimate the pathological complete response rate following neoadjuvant radiotherapy with concurrent capecitabine and oxaliplatin (CAPOX), with or without cetuximab based on the KRAS mutation status in rectal cancer.

Hypothesis: Cetuximab, a monoclonal antibody targeted against the EGF receptor, is active in metastatic colorectal cancer and a radio-sensitizer. In colorectal cancer, the presence of KRAS mutation has been associated with the absence of response to cetuximab. We hypothesise that the addition of cetuximab to CAPOX concurrent with neoadjuvant radiotherapy only benefited patients whose tumours do not have the KRAS mutation and therefore, personalizing cetuximab therapy based on tumour KRAS mutation status may yield a higher pathological response.

Methods: This study employed a standard 2-stage Phase II design to evaluate the efficacy and tolerability of two neoadjuvant chemoradiotherapy regimens. The assignment of the neoadjuvant chemotherapy will be determined by the KRAS mutation status of the tumor. Subjects with KRAS mutation will receive CAPOX. Subjects with no KRAS mutation will be randomized to receive CAPOX +/- cetuximab.Definitive surgery is scheduled for 6-8 weeks after the completion of chemoradiotherapy. Surgical management will be a sphincter preservation approach whenever possible, using the total mesorectal excision technique.After the operation, pathologic evaluation of the surgical specimen will be performed.

Significance:In this proof-of-concept study, we aim to demonstrate that using an enriched patient cohort to test our hypothesis that the addition of cetuximab will yield a higher pathological response rate in KRAS mutation-negative rectal cancer. This approach can potentially identify a subset of patients that may benefit from cetuximab and spare those who may not benefit from unnecessary treatment toxicities and costs. Our study will help to prioritise novel targeted agents for a smaller, faster, and less expensive confirmatory phase III trials.

ELIGIBILITY:
Inclusion Criteria:

1. All patients must have histologically or cytologically confirmed T3/4 and/or node positive adenocarcinoma of the rectum with the inferior border within 12 cm from the anal verge without evidence of distant metastases, as evaluated by computed tomography, ultrasonography, MRI or clinically.
2. Patients must have normal organ and marrow function as defined below:

   leukocytes >3,000/mcL absolute neutrophil count >1,500/mcL platelets >100,000/mcL total bilirubin within normal institutional limits AST(SGOT)/ALT(SGPT) greater than 2.5 X institutional upper limit of normal creatinine within normal institutional limits
3. Age >21 years
4. Patients must have ECOG performance status of 0-2.
5. Patients must be 18 years old or greater.
6. The tumor must be considered by the surgeon to be amenable to curative resection.
7. Ability to understand and the willingness to sign a written informed consent document.
8. Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

Exclusion Criteria:

1. Patients who have had prior chemotherapy or radiotherapy.
2. Patients may not be receiving any other investigational agents.
3. Patients with stage I or IV cancer of the rectum.
4. History of allergic reactions attributed to compounds of similar chemical or biologic composition to cetuximab, oxaliplatin or capecitabine.
5. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
6. Inability to take oral medications.
7. Pregnant women are excluded from this study because agents use in the study may cause fetal harm.
8. HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with docetaxel. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy.
9. History of other malignancies within 5 years, except non-melanoma skin cancer, in situ carcinoma of the cervix or ductal carcinoma of the breast. Previous invasive cancer permitted if disease-free at least 5 years.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74
Dates: Start 2008-07; Primary Completion 2014-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Wei Peng Yong, MRCP, MB ChB, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore

REFERENCES:
- [Background] Lievre A, Bachet JB, Le Corre D, Boige V, Landi B, Emile JF, Cote JF, Tomasic G, Penna C, Ducreux M, Rougier P, Penault-Llorca F, Laurent-Puig P. KRAS mutation status is predictive of response to cetuximab therapy in colorectal cancer. Cancer Res. 2006 Apr 15;66(8):3992-5. doi: 10.1158/0008-5472.CAN-06-0191. PMID 16618717
- [Background] Sauer R, Becker H, Hohenberger W, Rodel C, Wittekind C, Fietkau R, Martus P, Tschmelitsch J, Hager E, Hess CF, Karstens JH, Liersch T, Schmidberger H, Raab R; German Rectal Cancer Study Group. Preoperative versus postoperative chemoradiotherapy for rectal cancer. N Engl J Med. 2004 Oct 21;351(17):1731-40. doi: 10.1056/NEJMoa040694. PMID 15496622